CLINICAL TRIAL: NCT01709487
Title: Feasibility Study of Hyperthermic Intraperitoneal Chemotherapy (HIPEC) for Patients With Stage III or Only Pleural Stage IV Ovarian Carcinoma in First Line Therapy
Brief Title: Feasibility Study of HIPEC for Patients With Stage III or Only Pleural Stage IV Ovarian Carcinoma in First Line Therapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIPEC
Record Dates: First submitted 2012-10-12; First posted 2012-10-18 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2014-07

CONDITIONS: Ovarian Carcinoma; Fallopian Tube Carcinoma; Primary Peritoneal Carcinoma
Keywords: HIPEC; ovarian carcinoma; Bordet
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HIPEC surgery with chemotherapy (Experimental): * 3 courses of pre-operative chemotherapy: carboplatin AUC = 5 IV + paclitaxel 175 mg/m2 IV every 3 weeks
  * Debulking surgery
  * HIPEC with cisplatin 50 mg/m2 intraperitoneally at the end of surgery
  * 3 courses of post-operative chemotherapy: carboplatin AUC = 5 IV + paclitaxel 175 mg/m2 IV every 3 weeks
  Interventions: Procedure: HIPEC

INTERVENTIONS:
Procedure: HIPEC — HIPEC with cisplatin 50 mg/m2 intraperitoneally at the end of surgery

SUMMARY:
First line treatment for advanced ovarian carcinoma hyperthermic intraperitoneal chemotherapy (HIPEC) after optimal debulking.

DETAILED DESCRIPTION:
Addition of HIPEC to the standard first line treatment of ovarian carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* stage III or only pleural stage IV ovarian carcinoma first line treatment

Exclusion Criteria:

* incomplete surgery poor performance status bad general condition

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
mortality rate | 24 weeks
  We will record the mortality rate of our interventions: 3 cycles of pre-operative chemotherapy, surgery and HIPEC, 3 cycles of post-operative chemotherapy.

SECONDARY OUTCOMES:
progression free survival | 3 years
Overall survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Kerger, M.D., Principal Investigator — Institut Jules Bordet, Brussels, Belgium.; Frédéric Goffin, M.D., Principal Investigator — Hopital de la Citadelle, Liège, Belgium.
Locations (2):
- Belgium (2):
  - Hopital de la Citadelle, Liège, Liège
  - Institut Jules Bordet, Brussels